CLINICAL TRIAL: NCT02443714
Title: Pharmacokinetic and Pharmacodynamic Profile of Insulin Lispro Using Needle-Free Jet Injection Technology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor, Chongqing Medical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NFJI-2015
Record Dates: First submitted 2015-05-01; First posted 2015-05-14 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Needle-Free Jet Injection; Insulin Lispro; pharmacokinetics; pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Needle-free jet injection (Experimental): Jet injectors deliver insulin at a high velocity (typically.100 m/s) across the skin in the subcutaneous tissue and may dispense the insulin over a larger area than insulin injected with a syringe.
  Interventions: Device: Needle-free jet injection with insulin lispro
- Conventional pen (Experimental): Conventional insulin administration with insulin pens.
  Interventions: Device: Conventional pen injection with insulin lispro

INTERVENTIONS:
Device: Needle-free jet injection with insulin lispro — Subjects injected by jet injectors which deliver insulin lispro
  Arms: Needle-free jet injection
Device: Conventional pen injection with insulin lispro — Subjects injected by conventional insulin pens which deliver insulin lispro
  Arms: Conventional pen

SUMMARY:
Needle-free jet injector provides an alternative for patients with diabetes treated by insulin. This study aimed at evaluating pharmacokinetics and pharmacodynamics (PK-PD) profiles of lispro administered by jet injector and conventional pen.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, crossover study. Eighteen healthy volunteers will be recruited. Lispro (0.2 units/kg) will be administered by jet injector or by conventional pen and a seven-hour euglycemic clamp test will be performed. PK-PD profiles of lispro will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. The range of height should be 170±10cm.
2. The range of weight should be ±10%kg.
3. Liver and renal function should be normal.
4. Health subjects with no chronic diseases or medications.

Exclusion Criteria:

1. Drug allergy, history of allergic disorders or allergies.
2. A history of liver or kidney disease.
3. Smoker, drinkers.
4. Subjects who participated in other drug trials within a month.
5. Subjects who used medication which is known to organ damage.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Early insulin exposure | The area under the curve (AUC) of insulin from 0 to 30min (AUCins, 0-30min)

SECONDARY OUTCOMES:
Pharmacodynamics | AUC of GIR for 0-30 min, 30-60 min, 60-90 min, 90-120 min, 0-420 min,respectively
Pharmacodynamics | 50% glucose clearance time (GIR- TAUC50%)
Pharmacodynamics | Time to maximum GIR (GIR-Tmax)
Pharmacodynamics | Maximum GIR (GIRmax)
Pharmacokinetics | AUC of insulin concentration for 30-60 min, 60-90 min, 90-120 min, 0-420 min,respectively
Pharmacokinetics | The time to peak plasma insulin concentrations (Ins-Tmax)
Pharmacokinetics | The maximal insulin levels (Ins-Cmax)
Pharmacokinetics | 50% insulin absorption time (Ins-TAUC50%)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Sarno MJ, Bell J, Edelman SV. Pharmacokinetics and glucodynamics of rapid-, short-, and intermediate-acting insulins: comparison of jet injection to needle syringe. Diabetes Technol Ther. 2002;4(6):863-6. doi: 10.1089/152091502321118865. No abstract available. PMID 12614490
- [Result] Engwerda EE, Tack CJ, de Galan BE. Needle-free jet injection of rapid-acting insulin improves early postprandial glucose control in patients with diabetes. Diabetes Care. 2013 Nov;36(11):3436-41. doi: 10.2337/dc13-0492. Epub 2013 Oct 2. PMID 24089542
- [Result] Engwerda EE, Abbink EJ, Tack CJ, de Galan BE. Improved pharmacokinetic and pharmacodynamic profile of rapid-acting insulin using needle-free jet injection technology. Diabetes Care. 2011 Aug;34(8):1804-8. doi: 10.2337/dc11-0182. Epub 2011 Jun 29. PMID 21715522